CLINICAL TRIAL: NCT05901402
Title: Application of Aerobic and Resistance Exercise in Blood Glucose Control in Pregnant Women With GDM.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2023-07-102
Record Dates: First submitted 2023-04-24; First posted 2023-06-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Aerobic and Resistance Exercise
Keywords: the pregnant women with GDM; blood glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The experimental group performed aerobic resistance exercise during pregnancy every day.
  Interventions: Behavioral: aerobic and resistance exercise
- The control group (No Intervention): The control group was given traditional nursing.

INTERVENTIONS:
Behavioral: aerobic and resistance exercise — The experimental group performed aerobic resistance exercise during pregnancy every day.
  Arms: The experimental group

SUMMARY:
Objective:The aim of this study was to explore the rationality and clinical value of aerobic exercise during pregnancy in blood glucose control of pregnant women with GDM, and to provide theoretical basis for more appropriate clinical exercise management.

Method:The subjects of gestational diabetes in the hospital from March 2023 to May 2024 were studied. The exercise exercise with daily responsible nurses was based on resistance exercise, mainly with upper limb muscle exercise, supplemented by lower limb muscle exercise and aerobic exercise. Fasting blood glucose, 2 hours postprandial blood glucose and HbA1c in pregnant women with GDM were monitored.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with GDM without contraindications.
* Pregnant women with GDM who volunteered to participate in the project.
* Pregnant women give informed consent.

Exclusion Criteria:

* Pregnant women give up voluntarily.
* Hypoglycemia: In the presence of dizziness and other uncomfortable symptoms, people should stop exercising immediately, monitor blood sugar, and always prepare candy.
* Abdominal pain, vaginal bleeding and other symptoms of contraction should stop exercising immediately and seek medical attention in time.
* Fall: It is recommended to ensure the safety of the sports ground before exercise: keep the ground dry, clean, not easy to slip, no debris; Comfortable clothing and non-slip exercise are recommended.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | Collect blood samples and monitor fasting blood glucose in pregnant womendaily until delivery, it can be monitored for up to 10 months.
  Fasting blood glucose in pregnant women with GDM
2 hours blood glucose | Collect blood samples and monitor 2 hours postprandial blood glucosedaily until delivery, it can be monitored for up to 10 months.
  2 hours postprandial blood glucose in pregnant women with GDM
HbA1c | Collect blood samples and monitor monthly until delivery, it can be monitored for up to 10 months.
  HbA1c in pregnant women with GDM
Maternal weight gain | Monitor weight daily until delivery by weighing scale, it can be monitored for up to 10 months.
  Maternal Weight Gain during Pregnancy
Pulse | Monitor the pulse of pregnant women in the experimental group during exercise until delivery, it can be monitored for up to 10 months.
  The pulse of pregnant women in the experimental group during exercise

CONTACTS AND LOCATIONS:
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China